CLINICAL TRIAL: NCT06230913
Title: Comparative Effects of Kinesiotaping Versus Pressure Garments on Secondary Upper Extremity Lymphedema Following Microsurgical Breast Reconstruction After Severe Chest Burns.
Brief Title: Kinesiotaping Versus Pressure Garments on Secondary Upper Extremity Lymphedema.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Gopal Nambi, Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHPT/023/01
Record Dates: First submitted 2023-12-23; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Lymphedema of Upper Arm; Burns Chest Right Lateral; Burns Chest Left Lateral
Keywords: Kinesiotaping; Pressure garments; Lymphedema; Chest burns; Breast reconstruction
MeSH Terms: conditions — Lymphedema | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping group (Experimental): To perform taping of the chest, the patient was asked to stand upright with the affected shoulder rotated externally. Five straps of the fan shaped tape were extended to the chest toward the affected axilla with 15% to 20% tension, and the anchor was positioned without tension in the anterior axilla on the sound side.
  Interventions: Device: Kinesiotape
- Pressure garment group (Active Comparator): The skin was washed and dried before applying the PG. The Premium Lymphedema Gradient Garment (Jobskin, Long Eaton, England) was used to apply PGs. This garment has a pressure gradient built into it, applying between 20 and 60 mm Hg for at least 15 to 18 hours each day for three weeks. The gradient counter pressure is applied using a gram tension.
  Interventions: Device: Pressure garment

INTERVENTIONS:
Device: Kinesiotape — To perform taping of the chest, the patient was asked to stand upright with the affected shoulder rotated externally. Five straps of the fan shaped tape were extended to the chest toward the affected axilla with 15% to 20% tension, and the anchor was positioned without tension in the anterior axilla on the sound side.
  Arms: Kinesiotaping group
Device: Pressure garment — The skin was washed and dried before applying the PG. The Premium Lymphedema Gradient Garment (Jobskin, Long Eaton, England) was used to apply PGs. This garment has a pressure gradient built into it, applying between 20 and 60 mm Hg for at least 15 to 18 hours each day for three weeks. The gradient counter pressure is applied using a gram tension.
  Arms: Pressure garment group

SUMMARY:
The goal of this randomised control study is to compare kinesiotaping and pressue garments in secondary upper extremity lymphedema following microsurgical breast reconstruction after severe chest burns.

The primary objective of this study was to compare the effects of kinesiotaping and pressure garments on limb circumference, handgrip strength, shoulder pain and disability index (SPADI), and limb circumference in patients with lymphedema following breast reconstruction due to chest burns.

The participants were randomly assigned to one of two groups: the kinesiotaping group (n = 28) and the pressure garments group (n = 28).

To perform taping of the chest in the kinesiotaping group, the patient was asked to stand upright with the affected shoulder rotated externally. Five straps of the fan-shaped tape were extended to the chest toward the affected axilla with 15% to 20% tension, and the anchor was positioned without tension in the anterior axilla on the sound side.

In the pressure garment group, the participant's skin was washed and dried before applying the PG. The Premium Lymphedema Gradient Garment (Jobskin, Long Eaton, England) was used to apply PGs. This garment has a pressure gradient built into it, applying between 20 and 60 mm Hg for at least 15 to 18 hours each day for three weeks.

DETAILED DESCRIPTION:
The participants were randomly assigned to one of two groups: the kinesiotaping group (n = 28) and the pressure garments group (n = 28).

To perform taping of the chest in the kinesiotaping group, the patient was asked to stand upright with the affected shoulder rotated externally. Five straps of the fan-shaped tape were extended to the chest toward the affected axilla with 15% to 20% tension, and the anchor was positioned without tension in the anterior axilla on the sound side.

In the pressure garment group, the participant's skin was washed and dried before applying the PG. The Premium Lymphedema Gradient Garment (Jobskin, Long Eaton, England) was used to apply PGs. This garment has a pressure gradient built into it, applying between 20 and 60 mm Hg for at least 15 to 18 hours each day for three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Microsurgical breast reconstruction after severe chest burns.
* the patient's arm circumference should be at least more than 2cm but not greater than 8 cm when compared to the same site on the opposite arm.

Exclusion Criteria:

* Conditions that resulted in oedema or swelling,
* medication like diuretics,
* infections,
* allergies,
* other systemic diseases,
* pregnancy,
* bilateral lymphadenitis

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Microsurgical breast reconstruction after severe chest burns.
Enrollment: 56 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Arm circumference: | Baseline
  To measure the arm circumference, the patient lays in a prone position with their arms relaxed by the side of the body. A measuring tape is used to take the measurement. It was measured starting with 3 cm on the ulnar styloid process and proceeding with 45 cm proximal, and additionally at the metacarpal bones and midhand. For an accurate reading, the tape was snugly wrapped around the arm. The measurements were recorded for both the affected and unaffected arms, and the difference between the two measurements was then recorded under the title "circumference difference"
Arm circumference: | 2 months
  To measure the arm circumference, the patient lays in a prone position with their arms relaxed by the side of the body. A measuring tape is used to take the measurement. It was measured starting with 3 cm on the ulnar styloid process and proceeding with 45 cm proximal, and additionally at the metacarpal bones and midhand. For an accurate reading, the tape was snugly wrapped around the arm. The measurements were recorded for both the affected and unaffected arms, and the difference between the two measurements was then recorded under the title "circumference difference"
Arm circumference: | 6 months
  To measure the arm circumference, the patient lays in a prone position with their arms relaxed by the side of the body. A measuring tape is used to take the measurement. It was measured starting with 3 cm on the ulnar styloid process and proceeding with 45 cm proximal, and additionally at the metacarpal bones and midhand. For an accurate reading, the tape was snugly wrapped around the arm. The measurements were recorded for both the affected and unaffected arms, and the difference between the two measurements was then recorded under the title "circumference difference"
Arm circumference: | 12 months
  To measure the arm circumference, the patient lays in a prone position with their arms relaxed by the side of the body. A measuring tape is used to take the measurement. It was measured starting with 3 cm on the ulnar styloid process and proceeding with 45 cm proximal, and additionally at the metacarpal bones and midhand. For an accurate reading, the tape was snugly wrapped around the arm. The measurements were recorded for both the affected and unaffected arms, and the difference between the two measurements was then recorded under the title "circumference difference"

SECONDARY OUTCOMES:
Functional disability - SPADI | Baseline
  It is a tool to measure shoulder pain and disability. It consists of 13 criterias to assess pain and disabilty: 5 criterias assess pain and 8 assess disability. The reliability of its coefficients is ICC ≥0.89 and has shown high internal consistency.
Functional disability - SPADI | 2 months
  It is a tool to measure shoulder pain and disability. It consists of 13 criterias to assess pain and disabilty: 5 criterias assess pain and 8 assess disability. The reliability of its coefficients is ICC ≥0.89 and has shown high internal consistency.
Functional disability - SPADI | 6 months
  It is a tool to measure shoulder pain and disability. It consists of 13 criterias to assess pain and disabilty: 5 criterias assess pain and 8 assess disability. The reliability of its coefficients is ICC ≥0.89 and has shown high internal consistency.
Functional disability - SPADI | 12 months
  It is a tool to measure shoulder pain and disability. It consists of 13 criterias to assess pain and disabilty: 5 criterias assess pain and 8 assess disability. The reliability of its coefficients is ICC ≥0.89 and has shown high internal consistency.
Handgrip strength | Baseline
  a handheld dynamometer (78010, Lafayette Instrument Company, Loughboroug, Leics, England) was used to measure the hand grip strength. To record the hand grip strength, the patient is positioned in the standing position with their shoulder adducted, elbows flexed at an angle of 90 degrees with the forearm in mid position. The patient is asked to grip the device to the maximum of his capacity, the average of 3 readings are recorded.
Handgrip strength | 2 months
  a handheld dynamometer (78010, Lafayette Instrument Company, Loughboroug, Leics, England) was used to measure the hand grip strength. To record the hand grip strength, the patient is positioned in the standing position with their shoulder adducted, elbows flexed at an angle of 90 degrees with the forearm in mid position. The patient is asked to grip the device to the maximum of his capacity, the average of 3 readings are recorded.
Handgrip strength | 6 months
  a handheld dynamometer (78010, Lafayette Instrument Company, Loughboroug, Leics, England) was used to measure the hand grip strength. To record the hand grip strength, the patient is positioned in the standing position with their shoulder adducted, elbows flexed at an angle of 90 degrees with the forearm in mid position. The patient is asked to grip the device to the maximum of his capacity, the average of 3 readings are recorded.
Handgrip strength | 12 months
  a handheld dynamometer (78010, Lafayette Instrument Company, Loughboroug, Leics, England) was used to measure the hand grip strength. To record the hand grip strength, the patient is positioned in the standing position with their shoulder adducted, elbows flexed at an angle of 90 degrees with the forearm in mid position. The patient is asked to grip the device to the maximum of his capacity, the average of 3 readings are recorded.
QOL | Baseline
  The was assessed by cancer-specific questionnaire (EORTC QLQ-C30). It is composed of 30 questions, including functional scores (physical, social, emotional, and cognitive aspects). The functional scores ranged between 0 and 100, and higher scores indicated better condition. This questionnaire also included symptoms score (pain, dyspnea, fatigue, insomnia, nausea, loss of appetite, and financial problems). The symptom scores ranged from 100 to 0, and lower scores indicated better condition.
QOL | 2 months
  The was assessed by cancer-specific questionnaire (EORTC QLQ-C30). It is composed of 30 questions, including functional scores (physical, social, emotional, and cognitive aspects). The functional scores ranged between 0 and 100, and higher scores indicated better condition. This questionnaire also included symptoms score (pain, dyspnea, fatigue, insomnia, nausea, loss of appetite, and financial problems). The symptom scores ranged from 100 to 0, and lower scores indicated better condition.
QOL | 6 months
  The was assessed by cancer-specific questionnaire (EORTC QLQ-C30). It is composed of 30 questions, including functional scores (physical, social, emotional, and cognitive aspects). The functional scores ranged between 0 and 100, and higher scores indicated better condition. This questionnaire also included symptoms score (pain, dyspnea, fatigue, insomnia, nausea, loss of appetite, and financial problems). The symptom scores ranged from 100 to 0, and lower scores indicated better condition.
QOL | 12 months
  The was assessed by cancer-specific questionnaire (EORTC QLQ-C30). It is composed of 30 questions, including functional scores (physical, social, emotional, and cognitive aspects). The functional scores ranged between 0 and 100, and higher scores indicated better condition. This questionnaire also included symptoms score (pain, dyspnea, fatigue, insomnia, nausea, loss of appetite, and financial problems). The symptom scores ranged from 100 to 0, and lower scores indicated better condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Gopal Nambi, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data can be obtained by contacting the primary author.

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-12-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT06230913/SAP_000.pdf